CLINICAL TRIAL: NCT01983059
Title: A Multicenter Prospective Observational Cohort Study
Brief Title: Swiss Liver Venous Thrombosis Study
Acronym: SLVTS-SASL-35
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Other Study IDs: SLVTS-SASL-35
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, serum, plasma, stool and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Liver Venous Thrombosis

SUMMARY:
The Liver Venous Thrombosis Study is a prospective observational cohort study aimed at collecting clinical data, patient reported outcomes and biological samples of all patients who have been newly and previously diagnosed with liver venous thrombosis in one of the participating hospitals in- and out-patient clinics of the participating centers in Switzerland. All new patients diagnosed with liver venous thrombosis or patients who are currently being treated in one of the participating centers, will be asked to participate in the study.

DETAILED DESCRIPTION:
Background

Outcome measures:

Primary: Liver venous thrombosis recanalization

Secondary: Thrombosis progression, Overall mortality, Major bleeding, Ascites

Objective

* To start a prospective observational cohort study of Liver Venous Thrombosis patients in Switzerland from their primary diagnosis and already diagnosed patients.
* To examine long-term medical outcomes in patients with liver venous thrombosis in Switzerland by defining incidence, risk factors and treatment results
* To prospectively collect data on medical history, serious comorbidities, baseline clinical parameters, imaging results, pathology results, tumor characteristics, treatment, treatment outcomes, hospital stays, interventions and complications.
* To store in a biobank blood and biological samples, obtained during routine practice

Methods

N/A

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted in hospital or attend outpatient clinic
* Objectively confirmed portal vein thrombosis and/or hepatic vein thrombosis
* Budd-Chiari-Syndrome (BCS), Non-Cirrhotic Intrahepatic Portal Hypertension (NCIPH), Sinusoidal Obstructive Syndrome (SOS), Other Vascular Diseases (Hepatoportal Sclerosis (HC), Nodular Regenerative Hyperplasia (NRH), Obliterative Portal Venopathy (OPV) or Idiopathic Portal Hypertension (IPH))
* Subjects willing to provide informed consent

Exclusion Criteria

* Thrombosis limited to mesenteric or splenic vein
* Inability to sign consent form
* Follow-up not possible
* Cardiovascular, tumoral, pulmonary comorbidity with life expectancy estimated to be less than 6 months
* Portal vein invasion by hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Liver Venous Thrombosis patients in participating hospitals in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with liver venous thrombosis recanalization | End of study, expected to be on average after 5 years

SECONDARY OUTCOMES:
Number of patient with thrombosis recurrence and progression | End of study, expected to be on average after 5 years
Overall mortality | End of study, expected to be on average after 5 years
Number of patients with major bleeding | End of study, expected to be on average after 5 years
Number of patients with ascites | End of study, expected to be on average after 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Gottardi, Prof. Dr. med., Principal Investigator — Inselspital (University Hospital) Bern
Locations (8):
- Switzerland (8):
  - Department of Clinical Research, Hepatology Research Group, Bern, Canton of Bern
  - Klinik für Gastroenterologie und Hepatologie, Universtätsspital Basel, Basel, Kanton Basel
  - Medizinische Klinik - Kantonsspital Baden, Baden
  - Service de Gastro-entérologie et Hépatologie, Hôpitaux Universtaires de Genève, Geneva
  - Service de Gastroentérologie et d'Hépatologie, Centre Hospitalier Universitaire Vaudois, Lausanne
  - Centro di Epatologia - Clinica Luganese Moncucco, Lugano
  - Klinik für Gastroenterologie/Hepatologie, Kantonsspital St. Gallen, Sankt Gallen
  - Klinik für Gastroenterologie und Hepatologie Universitätsspital Zürich, Zurich